CLINICAL TRIAL: NCT06572098
Title: The Effect of Complex Decongestıve Therapy on Oxıdatıve Stress and Antıoxıdants In Patıents Wıth Lymphedema After Breast Cancer Treatment
Brief Title: The Effect of Complex Decongestıve Therapy on Oxıdatıve Stress and Antıoxıdants
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PDANALAN1
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: What Are the Effects of Lymphedema Treatment
Keywords: Breast cancer; Lymphedema; Oxidative stress
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Intervention Model Description: 1. Working Group (Complex decongestive therapy)
  2. Control Group
Who Masked: Participant
Masking Description: 1. Study Group-Patient with Lymphedema
  2. Control Group-Healthy Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- working group (Active Comparator): Patients will receive ten sessions of complex decongestive therapy. Patients will be evaluated for oxidative stress and antioxidant levels in three stages: before treatment, immediately after treatment and one month after the end of treatment.
  Interventions: Other: Complex decongestive therapy
- control group (No Intervention): As an evaluation parameter, a healthy female control group will be formed at least as many as the number of patients with lymphedema included in the study.

INTERVENTIONS:
Other: Complex decongestive therapy — Complex decongestive therapy consists of 4 phases. It will be performed by a lymphedema physiotherapist trained in Complex Decongestive Physiotherapy. Complex decongestive therapy consists of manual lymph drainage, skin care, multilayer bandaging and therapeutic exercises.
  Arms: working group

SUMMARY:
It is aimed to determine the changes of complex decongestive therapy applications on oxidative stress parameters and antioxidants in patients with lymphedema after breast cancer treatment.

DETAILED DESCRIPTION:
Lymphedema, which is the most common late complication of patients undergoing cancer treatment, affects the physical, social and psychological lives of the individual and decreases the quality of life as it causes motor dysfunctions, cosmetic deformations and psychological disorders. The addition of radiotherapy to surgical intervention increases the risk of lymphedema by 36%.

When free radicals increase in intensity, they cause structural defects in lipids, proteins and nucleic acids, and as a result, they are a cause and risk factor for chronic diseases such as cancer, neurodegenerative diseases and cardiovascular diseases.

Cancer cells produce high levels of reactive oxygen species (ROS) due to their fast metabolism and impaired cellular signaling mechanisms. High levels of ROS are generally harmful to cells and the redox state of cancer cells is different from normal cells. Therefore, cancer cells maintain ROS levels at a moderately high tumorigenic level, above the low cytostatic level, but below levels that may be cytotoxic. The oxidative stress state in a cancer cell is different from the oxidative stress state in a normal cell. It is also well known that increased oxidative stress and inflammation are associated with cancer risk. The number of studies investigating the effect of complex decongestive therapy, which is stated to be the most effective treatment method in the treatment of lymphedema, the most common complication after breast cancer treatment, on oxidative stress and antioxidant levels is quite limited.

In this study, it was aimed to reveal the changes of complex decongestive therapy applications on oxidative stress parameters and antioxidants in participants with lymphedema after breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Development of lymphedema after breast cancer treatment
* Clinical stage of lymphedema Stage-2 or Stage-3 diagnosis

Exclusion Criteria:

* Receiving treatment for lymphedema in the last three months
* Those diagnosed with severe heart failure and/or arrhythmia
* Persistent infection in the affected extremities
* Ongoing chemotherapy treatment
* Diagnosed with liver disease

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 52 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2027-04-03 (Estimated); Study Completion 2028-04-03 (Estimated)

PRIMARY OUTCOMES:
PON1 | will be assessed before treatment, immediately after treatment and one month after treatment.
  Paraoxonase

SECONDARY OUTCOMES:
OSİ | will be assessed before treatment, immediately after treatment and one month after treatment.
  Oxidative Stress Index

OTHER OUTCOMES:
LDL | will be assessed before treatment, immediately after treatment and one month after treatment.
  Low danditelilipoprotein
HDL | will be assessed before treatment, immediately after treatment and one month after treatment.
  High densitelilipoprotein
Trigliserit | will be assessed before treatment, immediately after treatment and one month after treatment.
  level of Trigliserit
GSH | will be assessed before treatment, immediately after treatment and one month after treatment.
  Rduktegulutathion
MDA | will be assessed before treatment, immediately after treatment and one month after treatment.
  malonDialdehyde

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Adana, çukurova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Toole J, Jammallo LS, Skolny MN, Miller CL, Elliott K, Specht MC, Taghian AG. Lymphedema following treatment for breast cancer: a new approach to an old problem. Crit Rev Oncol Hematol. 2013 Nov;88(2):437-46. doi: 10.1016/j.critrevonc.2013.05.001. Epub 2013 Jun 16. PMID 23777977
- [Background] Cormier JN, Askew RL, Mungovan KS, Xing Y, Ross MI, Armer JM. Lymphedema beyond breast cancer: a systematic review and meta-analysis of cancer-related secondary lymphedema. Cancer. 2010 Nov 15;116(22):5138-49. doi: 10.1002/cncr.25458. PMID 20665892